CLINICAL TRIAL: NCT02241694
Title: Haemophilia, Experiences, Results and Opportunities (HERO) in Brazil: Assessment of Psychological Effects of Haemophilia on Patients and Caregivers
Brief Title: To Quantify the Range of Main Psychosocial Factors Affecting Patients and Caregivers in Their Daily Lives
Acronym: HERO
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-4146; U1111-1147-4202 (Other: WHO)
Record Dates: First submitted 2014-09-01; First posted 2014-09-16 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors; Relatives to/Carers of Patients
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- survey
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given. Participants are to complete a questionnaire in the study.

SUMMARY:
This survey is conducted in South America. The purpose is to identify the key psychosocial issues affecting patients with haemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years or above with haemophilia A or B (with or without inhibitors) OR Parents/caregivers of children/adolescents younger than 18 years with haemophilia A or B (with or without inhibitors); only one subject per household will be able to participate
* Patients currently receiving one of the following treatments: a. replacement factor VIII therapy, b. replacement factor IX therapy, c. bypassing agents (recombinant factor VIIa or APCC) OR Patients with haemophilia, not receiving any kind of treatment with replacement factor VIII or IX or a bypassing agent (as appropriate), but who have had at least one spontaneous haemorrhage into one or more joints within the last 12 months
* The participants (patients with haemophilia and parents/caregivers for patients under 18 years old) must be able to complete a paper questionnaire in order to participate in the study
* Providing informed consent before the start of any study-related activities

Exclusion Criteria:

* Inability for the patients or parents/caregivers to understand and comply with verbal instructions, unless assisted by a member of the HTC (Haemophilia Treatment Center) or by a relative. (No other conditions were established for patients who cannot read or write to be able to participate in this study in addition to the need of help from a member of HTC or by a relative.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males with haemophilia and parents/carers of children with haemophilia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Qualitative assessments of perceived impact on daily life | Day 1

SECONDARY OUTCOMES:
Perceived disease control | Day 1
Carrier status and reactions to haemophilia diagnosis | Day 1
Genetic counselling and testing | Day 1
Impact of haemophilia in siblings | Day 1
Satisfaction with support from partners, family, friends, others | Day 1
Sexual intimacy with partners in long-term relationships | Day 1
Treatment method, compliance and location | Day 1
Modified WHO-5 (World Health Organization-Five Well Being Index) | Day 1
Knowledge and information about haemophilia | Day 1
Improvements in haemophilia care | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), GZZF, Study Director — Novo Nordisk A/S
Locations (1):
- Säo Paulo, Brazil

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com